CLINICAL TRIAL: NCT02088125
Title: Dynamic Ventilatory and Asymmetry of the Chest Wall During Breath Stacking and Volume-oriented Incentive Spirometer in Patients After Stroke: Crossover Clinical Trial
Brief Title: Dynamic Ventilatory and Asymmetry of the Chest Wall During Breath Stacking and Volume-oriented Incentive Spirometer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Catarina Souza Ferreira Rattes Lima, Dynamic ventilatory and asymmetry of the chest wall during breath stacking and volume-oriented incentive spirometer in patients after stroke: crossover clinical trial, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Stroke
Record Dates: First submitted 2014-02-24; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Stroke
Keywords: Stroke; Incentive Spirometry; Breath Stacking; Optoelectronic Plethysmography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incentive Spirometry (Active Comparator): The Incentive Spirometry was characterized by the use of the incentive spirometer volume, in which volunteer used a nasal clip and was instructed to inhale slowly and deeply through the mouthpiece of the equipment from functional residual capacity to total lung capacity.
  Interventions: Other: Incentive Spirometry
- Breath Stacking (Active Comparator): Breath Stacking A mask was used with two one-way valves (inspiratory limb and expiratory limb), which was coupled to the patient's face allowing only inspiration, while the expiratory branch remained occluded for the individual only perform successive inspiratory efforts.
  Interventions: Other: Breath Stacking

INTERVENTIONS:
Other: Breath Stacking — Breath Stacking A mask was used with two one-way valves (inspiratory limb and expiratory limb), which was coupled to the patient's face allowing only inspiration, while the expiratory branch remained occluded for the individual only perform successive inspiratory efforts.
  Arms: Breath Stacking
Other: Incentive Spirometry — The Incentive Spirometry was characterized by the use of the incentive spirometer volume, in which volunteer used a nasal clip and was instructed to inhale slowly and deeply through the mouthpiece of the equipment from functional residual capacity to total lung capacity.
  Arms: Incentive Spirometry

SUMMARY:
The purpose of the study was to analyze the effect of IS and BS on dynamics ventilatory and asymmetry of the chest wall in patients after stroke .

DETAILED DESCRIPTION:
All volunteers were undergone to two types of pulmonary expansion therapy (PET) techniques: volume incentive spirometry (VIS) and BS.

Procedures involved two distinct phases: assessment and intervention. In the first day was performed assessment of the participants to obtain the following data: anamnesis, initial evaluation using the Ashwouth Scale, Barthel Index and Mini Mental State Examination, anthropometric data and pulmonary function using spirometry and respiratory muscle pressures.

Intervention phase was performed in two different days, each day for only one PET techniques (VIS or BS), with a minimal wash-out period of one day according to the randomization sequence. Optoelectronic Pletysmography (OEP) was recorded during quite breathing at rest and during the execution of five maneuvers form each PET technique tested.

ELIGIBILITY:
Inclusion Criteria:Subjects with right hemiparesis due to stroke for more than three months, of both genders, most than 20 years, with scores between 1 and 3 for Ashworth Scale for upper limb, up to 85 for Index score Barthel and minimum score of 18 on the Mini Mental State Examination.

-

Exclusion Criteria: Facial paralysis, rheumatic or orthopedic diseases or deformities / abnormalities in the spine that could compromise the respiratory mechanics; reported respiratory conditions (asthma, chronic obstructive pulmonary disease, cystic fibrosis) or presenting spirometry with forced expiratory volume in one second (FEV1) below 80% predicted and compared VEF1/Capacitate Forced vital ≤ .7; history of recent abdominal or thoracic surgery and hemodynamic instability or pregnancy.

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Volume of the chest wall and Thoraco-abdominal compartments (pulmonary rib cage, abdominal rib cage and abdomen) | During assessment and intervention, on average for an hour
  Total chest wall and in the Differents thoraco-abdominal compartments measured by Opto-electronic plethysmography (OEP)

SECONDARY OUTCOMES:
Ventilatory Pattern (minute ventilation, breathing frequency, inspiratory time (TI), expiratory time (TE), duty cycle (TI/TTOT), tidal volume, mean inspiratory flow, mean expiratory flow) | During assessment and intervention, on average for an hour
  From variations of Volume of the chest wall during breathing measured by Opto-electronic plethysmography (OEP)

CONTACTS AND LOCATIONS:
Overall Officials: Armele Dornelas, PhD, Study Director — Federal University of Pernambuco Physiotherapy Department
Locations (1):
- Department of Physical Therapy, Federal University of Pernambuco, Recife, Pernambuco, Brazil, Recife, Pernambuco, Brazil